CLINICAL TRIAL: NCT02708368
Title: Investigation to Develop Standard Operating Procedures (SOP) for the Determination of Innovative CKD-MBD(Chronic Kidney Disease - Mineral Bone Disorder)-Serum-(Plasma-)Parameters
Brief Title: SOP's for CKD-MBD-Biomarkers
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: 15-109
Record Dates: First submitted 2016-02-29; First posted 2016-03-15 (Estimated); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Chronic Kidney Diseases
Keywords: Chronic Kidney Disease - Mineral Bone Disorder (CKD-MBD)
MeSH Terms: conditions — Renal Insufficiency, Chronic; Chronic Kidney Disease-Mineral and Bone Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients on dialysis: 16 patients on dialysis with a sex ratio 1:1; 8 patients on hemodialysis and 8 patients on hemodiafiltration
  Interventions: Other: blood withdrawal
- Healthy Subjects: 16 healthy subjects with a sex ratio 1:1
  Interventions: Other: blood withdrawal

INTERVENTIONS:
Other: blood withdrawal — 3 times

SUMMARY:
CKD-MBD (Chronic Kidney Disease - Mineral and Bone Disorder) is an extensive disease and includes dysfunction of the mineral metabolism, the bone metabolism and cardiovascular diseases in the context of renal insufficiency. Clinical pictures of peripheral artery occlusive disease (PAOD), Coronary artery disease (CAD) and arterial hypertension favours among other main risk factors (smoking, obesity, etc.) additional cardiovascular complications. For this reason it makes sense to monitor these patients regularly. For this purpose the determination of different biomarkers would be appropriate for control of the course of disease.

During various studies the biomarkers FGF23, s-klotho, sclerostin, DKK1, BMP2, YKL-40 und MGP were established as indicators for the disease activity, as diagnostic criteria for the existence of CKD-MBD or as risk markers for the incidence of adverse events (incl. death) within the scope of CKD-MBD. For the clinical routine care application of these parameters standard operating procedures (SOP) are missing for the determination method relating to optimal pre-analytic and analytic procedures. These analyses are necessary to ensure the reproducibility of study results and to transfer these parameters in the clinical daily routine for risk stratification.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are regularly (3 times a week) on dialysis in the Maria-Hilf-Clinic or healthy subjects
* Male or Female at the age of at least 18 years
* Patients who will be admitted to the clinics of the University Hospital RWTH Aachen or of the Maria-Hilf-Clinic Mönchengladbach or healthy subjects
* written informed consent form
* Subjects who are contractually capable and mentally able to understand and follow the instructions of the study personnel

Exclusion Criteria:

* age < 18 years
* subjects who are unwilling or not able to consent
* pregnant or lactating women
* subject has been committed to an institution by legal or regulatory order
* dependency or working relationship with the investigator
* participation in a parallel interventional clinical study
* Hb-value < 10 g/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who are regularly on dialysis in the clinics will be selected . Healthy Subjects will be recruited over notices in clinic.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2016-11-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
an optimal analysis of innovative CKD-MBD-Biomarkers | through study completion, an average of 3 months

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Department of Medicine, Division of Cardiology, Pulmonary Diseases and Vascular Medicine at the University Hospital, RWTH Aachen, Aachen, North Rhine-Westphalia
  - Clinic for Nephrology and Diabetology, Hospital St. Franziskus (Maria-Hilf-Clinic), Mönchengladbach, North Rhine-Westphalia

IPD SHARING:
Plan to Share IPD: No